CLINICAL TRIAL: NCT00943345
Title: Dubbelblind Crossover Study for Validation of New Tests for Gastrointestinal (GI) Permeability
Brief Title: Validation of New Tests for Gastrointestinal (GI) Permeability
Acronym: Permeability
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Kim van Wijck, MD, PhD student, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MEC 09-3-034
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Gastrointestinal Diseases
Keywords: GI; gastrointestinal; permeability; indometacin; indomethacin; coeliac
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GS dual sugar permeability test (Active Comparator): Golden standard GI permeability test - testing occurs for basal permeability (with placebo) and after ingestion of indometacin (for normal controls).
  Coeliac patients will only have 1 test to assess basal GI permeability.
  Interventions: Drug: indometacin
- Multi sugar test (Other): New GI permeability test - testing occurs for basal permeability (with placebo) and after ingestion of indometacin (for normal controls).
  Coeliac patients will only have 1 test to assess basal GI permeability.
  Interventions: Drug: indometacin
- Protein test (Other): New GI permeability test - testing occurs for basal permeability (with placebo) and after ingestion of indometacin (for normal controls).
  Coeliac patients will only have 1 test to assess basal GI permeability.
  Interventions: Drug: indometacin
- PEG test (Other): New GI permeability test - testing occurs for basal permeability (with placebo) and after ingestion of indometacin (for normal controls).
  Coeliac patients will only have 1 test to assess basal GI permeability.
  Interventions: Drug: indometacin

INTERVENTIONS:
Drug: indometacin — * capsule for oral consumption
  * at 22h00 evening before test day: 75 mg
  * at 7h30 on the test day: 50 mg This intervention will be applied 4 times (4 arms).
  Other Names: Indometacin [Actavis]

SUMMARY:
Introduction: The primary function of the gastrointestinal (GI) wall is digestion and absorption of nutrients that are important for growth and development. The second important function of the GI wall is forming an effective barrier to prevent penetration of potentially harmful components from the inside of the gut (lumen), via the GI wall, into the body.

A compromised barrier function may play an important role in the development of a range of inflammatory GI diseases such as coeliac disease, Inflammatory Bowel Disease (IBD), food allergy, but also in the pathophysiology of postoperative complications. It is important and clinically relevant to have reliable GI permeability tests, however the existing test leave room for improvement.

Rationale/aim: Three new tests are developed to assess gastrointestinal permeability in both normal controls with and without raised permeability, and in patients with coeliac disease. In the current study these new permeability tests will be evaluated and compared with the golden standard permeability test, the dual sugar test.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls, female/male, 18-75 years of age, OR:
* coeliac disease without taking medicine, female/male, 18-75 years of age

Exclusion Criteria:

* cardiac and/or vascular disease
* chronic obstructive pulmonary disease (COPD)
* rheumatic arthritis (RA)
* Inflammatory bowel disease(IBD); Crohn's colitis or colitis ulcerosa
* Irritable bowel syndrome (IBS)
* Inflammatory systemic disease
* Obesity (Body Mass Index ≥ 30 kg/m²)
* Diabetes Mellitus
* Thyroid disease
* Kidney disease
* Cancer
* Smoking
* Substance abuse (alcohol, drug, cocain, opioids, and others)
* Use of drugs
* Operations to the GI system, apart from appendectomy
* Allergy to eggs or milk
* Hypersensitivity to any of the following: lactulose, l-rhamnose, sucrose, sucralose of erythritol
* Acute porphyria or phenylketonuria (PKU)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of permeability tests (new versus golden standard dual sugar test) | 24 hours

SECONDARY OUTCOMES:
GI permeability | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: WA Buurman, Prof.dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Zuid-Limburg, Netherlands

REFERENCES:
- [Derived] van Wijck K, Verlinden TJ, van Eijk HM, Dekker J, Buurman WA, Dejong CH, Lenaerts K. Novel multi-sugar assay for site-specific gastrointestinal permeability analysis: a randomized controlled crossover trial. Clin Nutr. 2013 Apr;32(2):245-51. doi: 10.1016/j.clnu.2012.06.014. Epub 2012 Aug 11. PMID 22892368